CLINICAL TRIAL: NCT06227494
Title: Dietary Fiber: Is it the Missing Link in Achieving Long Term Behavior Change?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-59-STW
Record Dates: First submitted 2023-07-28; First posted 2024-01-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fiber Intervention (Experimental): Individuals in this arm will be given instruction on how to increase fiber intake,
  Interventions: Behavioral: Fiber Intervention
- Standard Weight Loss Education (Active Comparator): Individuals in this arm will be given standard weight loss education
  Interventions: Behavioral: Standard Weight Loss Education
- Fiber Intervention + Standard Weight Loss Education (Experimental): Individuals in this arm will be given education on both fiber and standard weight loss
  Interventions: Behavioral: Fiber Intervention; Behavioral: Standard Weight Loss Education

INTERVENTIONS:
Behavioral: Fiber Intervention — Group education and phone-based motivational interviewing to gradually increase dietary fiber consumption to 30-35 grams per day.
  Arms: Fiber Intervention; Fiber Intervention + Standard Weight Loss Education
Behavioral: Standard Weight Loss Education — Group education and phone-based motivational interviewing to promote current evidence-based behaviors to promote weight loss via achieving a negative energy balance.
  Arms: Fiber Intervention + Standard Weight Loss Education; Standard Weight Loss Education

SUMMARY:
The overall objective of this three-arm randomized controlled trial is to compare a dietary fiber-focused behavioral intervention to standard weight loss education for improving eating-related behavior and cognition, weight, and metabolic markers of chronic disease risk in a population of adults with obesity.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Dietary fiber intake ≤25 grams/day
* Self-reported BMI ≥30 kg/m2
* Willingness to attend in-person education sessions
* Willingness to avoid taking supplemental digestive aids (e.g., alpha-galactosidase (Beano®),
* Willingness to provide informed consent.

Exclusion Criteria:

* Metabolic, digestive, or allergic conditions or reactions that preclude consumption of whole food or food groups (e.g., irritable bowel syndrome, diverticulosis)
* History of gastric bypass surgery
* Currently taking glucagon like glucagon-like peptide-1 (GLP-1) Receptor Agonists
* Self-reported history of a diagnosed eating disorder
* Chronic disease (other than obesity)
* Pregnancy or lactation
* Use of tobacco or electronic smoking products
* Taking a pre-, pro-, or syn-biotic supplement
* Enrollment in another weight loss or diet intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Body weight | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Measure of body weight/mass

SECONDARY OUTCOMES:
Body composition (fat mass, lean mass) | Measured at baseline (time 1, month 0) and post-observation (time 3, month 27)
  Dual x-ray absorptiometry (DEXA) scans
Fecal short chain fatty acids | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Taken from fecal samples collected at home
Fecal bacteria measured using 16S ribosomal ribonucleic acid (rRNA) sequencing | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Will include measures of diversity, abundance, etc.
Total Cholesterol | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Measured via blood samples (unit= milligram/deciliter (mg/dL))
Fasting blood glucose | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 33, month 27)
  Measured via blood samples (unit=mg/dL)
Healthy Eating Index Scores measured using Health Eating Index 2020 (HEI-2020) | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Taken from 3 day diet records (score range=0-100, higher=better diet quality)
Three-Factor Eating Questionnaire | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Resulting scores in uncontrolled eating (range=9-36), cognitive restraint (range=3-12), and emotional eating (range=6-24); higher scores indicate more of that particular eating behavior
Implicit Association Test | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Represented with a total D variable (No range, but more negative = greater preference for unprocessed food)
Behavioral Inhibition System/Behavioral Approach System (BIS/BAS) Scale | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Score ranges from 20 to 80, with higher scores indicating greater behavioral inhibition and behavioral activation
Executive Function: Tower Test (Delis-Kaplan Executive Function System) | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Total Achievement Score (range=0-30, higher = higher executive function)
Executive Function: Color-Word Interference Test (Delis-Kaplan Executive Function System) | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Scaled inhibition/switching scores (score range=1-19, higher = higher executive function)
Skin Carotenoid scores measured via the Veggie Meter | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Veggie Meter; score range 0-800 (higher=greater skin carotenoids (i.e., consumption of more fruits/vegetables)
High-density lipoprotein (HDL) cholesterol | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Measured via blood samples (unit=mg/dL)
Low-density lipoprotein (LDL) cholesterol | Measured at baseline (time 1, month 0), post-intervention (time 2, month 15), and post-observation (time 3, month 27)
  Measured via blood samples (unit=mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No